CLINICAL TRIAL: NCT05040438
Title: A Phase 2a Study Using Natural Killer (NK) Cell Therapy Combined With Hepatic Artery Infusion Chemotherapy (HAIC) in Patients With Locally Advanced Hepatocellular Carcinoma
Brief Title: Natural Killer (NK) Cell Therapy in Locally Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxcell Bio, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vax-NK/HCC-201
Record Dates: First submitted 2021-08-26; First posted 2021-09-10 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-05

CONDITIONS: Locally Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous NK cell infusion combined with HAIC (Experimental): HAIC of 5-FU (500 mg/m2, Q4W) and cisplatin (15 mg/m2, Q4W) will be administered for up to 4 cycles to patients with locally advanced HCC. Subjects who achieved sustained SD or better based on the mRECIST criteria after 2nd cycle of HAIC will be enrolled to receive 1x10^9 cells VAX-NK/HCC infusion.
  Interventions: Biological: Vax-NK/HCC

INTERVENTIONS:
Biological: Vax-NK/HCC — autologous NK cells expanded ex vivo.

SUMMARY:
This Phase 2a trial will evaluate the safety and efficacy of NK cell therapy combined with the hepatic artery infusion chemotherapy (HAIC) in patients with intermediate and/or locally advanced hepatocellular carcinoma (HCC). We hypothesized that 5-fluorouracil (FU) with immunomodulatory functions would relieve the immunosuppressive microenvironment from the myeloid-derived suppressor cells (MDSCs), thereby enhancing the anti-tumor activity of NK cells. Thus, the subsequent infusion of autologous NK cells (VAX-NK/HCC) following HAIC treatment may further improve the anti-tumor activity in patients with advanced HCC.

DETAILED DESCRIPTION:
Primary Objective I. To assess the objective response rate (ORR) of administering VAX-NK/HCC, autologous NK cells combined with HAIC in patients with locally advanced HCC.

Secondary Objectives I. To assess the efficacy of administering VAX-NK/HCC combined with HAIC. II. To assess the safety of administering VAX-NK/HCC combined with HAIC. III. To assess the immune responses of administering VAX-NK/HCC combined with HAIC.

OUTLINE: This is a Phase 2a study. Patients receive HAIC treatment every 4 week for up to 4 cycles followed by ex-vivo expanded autologous NK cell infusions. The NK cell treatment repeats every 4 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients will be followed until the disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with intermediate and/or locally advanced HCC histologically confirmed by biopsy or by typical radiological findings.
* Subjects who were not suitable for or failed curative treatments such as surgical resection, local ablation therapy, transarterial chemoembolization (TACE), sorafenib, atezolizumab, bevacizumab, etc.
* Child-Pugh liver function class A or B.
* Subjects' ECOG performance status of 0 or 1.
* The presence of macrovascular invasion.
* Adequate liver, renal, and hematologic functions.

Exclusion Criteria:

* Subjects who received the immune cell-based therapy within 6 months before the screening visit.
* Subjects with a history of a malignancy other than HCC within the last 5 years, liver transplantation, and hypersensitivity to 5-FU or cisplatin.
* Subjects with extra-hepatic metastases.
* Subjects who have ongoing autoimmune disease.
* Female subjects who are pregnant or lactating or women of child-bearing potential but unable to take adequate contraception.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of administering VAX-NK/HCC combined with HAIC | average 6 months
  ORR will be measured as the proportion of patients with a best overall response of complete response (CR) and partial response (PR) of administering VAX-NK/HCC combined with HAIC.

SECONDARY OUTCOMES:
Disease control rate (DCR) of administering VAX-NK/HCC combined with HAIC | average 6 months
  ORR will be measured as the proportion of patients with a best overall response of complete response (CR), partial response (PR), and stable disease (SD) of administering VAX-NK/HCC combined with HAIC.
Time to progression (TTP) of administering VAX-NK/HCC combined with HAIC | average 6 months
  TTP will be measured by time to progression, defined as time from enrollment to disease progression.
Overall survival (OS) of administering VAX-NK/HCC combined with HAIC | average 12 months
  OS will be measured as time from enrollment to death due to any cause.
Quality of Life of administering VAX-NK/HCC combined with HAIC | average 6 months
  The assessment will be performed using the Korean versions of European Organization for Research and Treatment of Cancer (EORTC) Questionnaire 30 (QLQ-C30) consisting of 30 items. Total score: Range 0-100.
Adverse Events (AEs) and Serious Adverse Events (SAEs) of administering VAX-NK/HCC combined with HAIC | average 6 months
  The assessment will be measured by determining the number of patients that experience AEs and SAEs graded according to the NCI-CTCAE (Version 4.0)
The proportions of T and NK cells | average 6 months
  This will be measured by determining the relative percentages of CD4+CD8+ T cells and CD3- CD56+ NK cells in patients' peripheral blood.
The lymphocyte/monocyte ratio (LMR) | average 6 months
  LMR will be calculated by dividing the absolute lymphocyte count by the absolute monocyte count in patients' peripheral blood.
The NK cell cytotoxicity | average 6 months
  This will be measured by determining percent cell lysis of target cells (K562) in patients' peripheral blood.
The serum cytokine levels | average 6 months
  The serum concentrations of IFN-γ, IL-10, and TGF-β will be measured in patients' serum using the Enzyme-Linked immunosorbent assays.

CONTACTS AND LOCATIONS:
Overall Officials: Seon-Ah Ha, Ph.D., Study Director — VaxCell Biotherapeutics Co., Ltd.
Locations (1):
- Seon-Ah Ha, Hwasun, Jeollanam-do, South Korea